CLINICAL TRIAL: NCT01531855
Title: The Metabolic and Glycaemic Responses to Reductions in Rapid-acting Insulin Dose After Running Exercise in People With Type 1 Diabetes Mellitus.
Brief Title: Post-exercise Insulin Reductions in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: west-walker1
Record Dates: First submitted 2012-02-07; First posted 2012-02-13 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Type 1 Diabetes
Keywords: T1DM, Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin dose (Other): Reducing rapid-acting insulin dose (insulin aspart or lispro) after exercise.
  Interventions: Other: Reducing post-exercise rapid-acting insulin (insulin lispro or aspart) dose

INTERVENTIONS:
Other: Reducing post-exercise rapid-acting insulin (insulin lispro or aspart) dose — Dosage after exercise

SUMMARY:
The investigators hypothesise that reducing rapid-acting insulin dose after exercise will help prevent Type 1 diabetes individuals experiencing hypoglycaemia.

ELIGIBILITY:
Inclusion Criteria:

* T1DM,
* Male,
* basal-bolus regimen (insulin glargine / detemir with insulin lispro / aspart),
* HbA1c < 9.9%,
* aged 18-50.

Exclusion Criteria:

* HbA1c > 10%,
* not treated with basal-bolus (insulin glargine / detemir with insulin lispro / aspart),
* aged <18 > 50.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
24 hour blood glucose area under the curve | 24 hours
  24 hour, post-exercise, glucose area under the curve.

SECONDARY OUTCOMES:
Ketogenesis | 60 minutes before and 24 hours post-exercise
  Blood beta-hydroxybutyrate concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J West, Principal Investigator — Northumbria University
Locations (1):
- Clinical Research Facility, Newcaslte Upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Background] West DJ, Morton RD, Bain SC, Stephens JW, Bracken RM. Blood glucose responses to reductions in pre-exercise rapid-acting insulin for 24 h after running in individuals with type 1 diabetes. J Sports Sci. 2010 May;28(7):781-8. doi: 10.1080/02640411003734093. PMID 20496226
- [Derived] Campbell MD, Walker M, Trenell MI, Luzio S, Dunseath G, Tuner D, Bracken RM, Bain SC, Russell M, Stevenson EJ, West DJ. Metabolic implications when employing heavy pre- and post-exercise rapid-acting insulin reductions to prevent hypoglycaemia in type 1 diabetes patients: a randomised clinical trial. PLoS One. 2014 May 23;9(5):e97143. doi: 10.1371/journal.pone.0097143. eCollection 2014. PMID 24858952
- [Derived] Campbell MD, Walker M, Trenell MI, Jakovljevic DG, Stevenson EJ, Bracken RM, Bain SC, West DJ. Large pre- and postexercise rapid-acting insulin reductions preserve glycemia and prevent early- but not late-onset hypoglycemia in patients with type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2217-24. doi: 10.2337/dc12-2467. Epub 2013 Mar 20. PMID 23514728